CLINICAL TRIAL: NCT06764407
Title: The Effect of Patient Preferred Music on Postoperative Anxiety
Brief Title: The Effect of Music on Postoperative Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Burak NALBANT, assistant professor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 33
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Anxiety Postoperative; Quality of Recovery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient preferential music (Active Comparator): The preference of the patients will be listened to preoperatively through the headphones.
  Interventions: Other: Patient preferential music
- No Music (Placebo Comparator): Patients will not listen to music.
  Interventions: Other: No Music

INTERVENTIONS:
Other: Patient preferential music — Patients will listen to their preferred music through the headphones before surgery and intraoperative period.
  Arms: Patient preferential music
Other: No Music — Patients will not listen to music.
  Arms: No Music

SUMMARY:
In this study, it is planned to learned the effect of listening to the music preferred by the patient on postoperative anxiety.

DETAILED DESCRIPTION:
Preoperative anxiety can be detected via structured and standardized screening by the State-Trait Anxiety Inventory (STAI) I and II. 80 patients scheduled for total knee arthroplasty surgery for will be included in our study. Preoperative STAI I and II score (anxiety questionnaire) will be applied to each patient. The patients will be divided into two groups as listening patient preferential music, and control. The patient favorite music track and singer without limiting the kind of music or classical music will be played through the headphones.Secondary aim is to assess the effect of listening patient preferred music on Quality of recovery, postoperative pain, MCID (minimal clinically important diffirence), patient and surgeon satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Undergo Total Knee Arthroplasty Under Spinal Anesthesia

Exclusion Criteria:

* Poor vision
* Significant hearing loss
* Dementia
* Active opioid use
* Regular use of anxiolytics or discontinuation of them on the day of surgery
* Unwillingness to participate in the study
* Unwillingness to listening to music

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-01-09 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Spielberg State-Trait Anxiety Inventory (STAI) score | Preoperative 1st hour and Postoperative 4th hour
  The test scores between 20 and 80, with higher scores indicating more generalized and stronger anxiety. Preoperative and postoperative STAI I score questions will be asked.

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) | Postoperative 4th, 12th and 24th hours
  11-point numerical rating scale for pain (0='no pain' and 10='worst pain possible pain') were explained.
The quality of postoperative functional recovery (QoR-15) score | Preoperative 1st hour and Postoperative 24th hour
  The patient-reported Turkish QoR-15 score includes 15 questions that evaluate the patient's postoperative recovery. The QoR-15 score is grouped under two groups, A and B. A high QoR-15 score, a score between 0 (poor) and 10 (excellent) for each item, and a total score of 150 indicate better quality of recovery.
Patient satisfaction score | Postoperative 24th hour
  Patients were asked about their satisfaction levels with a number between 0-10.
MCID of STAI score | 24 hour
  Calculation of the MCID of the STAI score
MCID of QoR-15 score | 24 hour
  Calculation of the MCID of the QoR-15 score

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kavak Akelma F, Altinsoy S, Arslan MT, Ergil J. Effect of favorite music on postoperative anxiety and pain. Anaesthesist. 2020 Mar;69(3):198-204. doi: 10.1007/s00101-020-00731-8. Epub 2020 Feb 11. PMID 32047952
- [Background] Bradt J, Dileo C, Shim M. Music interventions for preoperative anxiety. Cochrane Database Syst Rev. 2013 Jun 6;2013(6):CD006908. doi: 10.1002/14651858.CD006908.pub2. PMID 23740695